CLINICAL TRIAL: NCT01837615
Title: Assessment of the Photopill Capsule Treatment for Safety and Feasibility in Patients With Ulcerative Proctitis
Brief Title: Assessment of Photopill Capsule Treatment for Safety and Feasibility in Ulcerative Proctitis
Acronym: Photopill
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Photopill Medical Ltd (Unknown)
Responsible Party: Principal Investigator, Hanke Brandse, MD, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL39583.018.12
Record Dates: First submitted 2013-04-18; First posted 2013-04-23 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2015-06

CONDITIONS: Ulcerative Colitis; Proctitis
Keywords: Ulcerative Colitis; Ulcerative Proctitis; Low Level Light Therapy; Safety; Efficacy
MeSH Terms: conditions — Colitis, Ulcerative; Proctitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Photopill treatment (Experimental)
  Interventions: Device: Photopill treatment

INTERVENTIONS:
Device: Photopill treatment
  Other Names: Photopill

SUMMARY:
Low Level Light therapy (LLLT) has been used for tissue healing in many mucosal diseases that involve wounds, ulcers and inflammation, oral chemotherapy-induced mucositis in particular. Likewise IBD is characterized by chronic tissue inflammation, tissue damage and ulcerations in various extents. Therefore we hypothesize that LLLT might be effective in treating IBD and the Photopill capsule was developed for this purpose.

An open-label, interventional, clinical trial was designed for assessment of the safety and feasibilty of the Photopill capsule treatment in patients with mild to moderate Ulcerative Proctitis.

Primary endpoints being: safety reflected by the number and severity of adverse events and mucosal appearance at sigmoidoscopies day 14, day 28, day 42 compared to baseline condition.

Furthermore clinical and biochemical parameters are monitored during the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Ulcerative Proctitis (Mayo grade 1/2)

Exclusion Criteria:

* Symptomatic hemorrhoids
* Pregnant or lactating females
* Patients that have used any experimental treatment within 8 weeks prior to Day 0
* Patient that have used any biologics therapies or immunomodulation agents and/or steroids 4 weeks prior to Day 0
* Rectal therapy 2 weeks prior to Day 0

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2013-01; Primary Completion 2015-05 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Adverse events | day 0-42
  Any adverse events reported by subjects

SECONDARY OUTCOMES:
Inflammatory markers | day 0,14,28,42
  serum CRP, serum Hb/Ht, fecal Calprotectin
Clinical Questionnaires | day 0,14,28,42
  Simple Clinical Colitis Activity Index Partial Mayo score
Mucosal appearance at sigmoidoscopy | week 0,14,28.42
  endoscopic disease activity Mayo score and possible damage by device

CONTACTS AND LOCATIONS:
Overall Officials: Geert R D'Haens, MD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Academic Medical Center, Amsterdam, North Holland, Netherlands